CLINICAL TRIAL: NCT06524882
Title: A Randomized Trial of Dichoptic Treatment for Amblyopia in Children 8 to 12 Years of Age
Brief Title: Dichoptic Treatment for Amblyopia in Children 8 to 12 Years of Age
Acronym: ATS24
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Pediatric Eye Disease Investigator Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS24; 2UG1EY011751 (NIH)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Amblyopia
Keywords: Dichoptic; Luminopia; Vivid Vision; Game; movie; glasses
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Luminopia Group (Experimental): dichoptic movies/shows wearing the Luminopia headset prescribed 1 hour per day (treatment time can be split into shorter sessions totaling 1 hour each day) 6 days a week with current optical correction if needed
  Interventions: Device: Luminopia
- Vivid Vision Group (Experimental): dichoptic games using the Vivid Vision headset, prescribed approximately 25 minutes per day (treatment time to complete the day's sessions can be split into shorter sessions totaling about 25 minutes each day) 6 days per week with current optical correction if needed
  Interventions: Device: Vivid Vision
- Continued Optical Correction Group (Active Comparator): continued full-time optical correction alone if needed
  Interventions: Device: Optical Correction

INTERVENTIONS:
Device: Vivid Vision — dichoptic video games played through a virtual reality headset
  Arms: Vivid Vision Group
Device: Luminopia — dichoptic movies/shows shown through a virtual reality headset
  Arms: Luminopia Group
Device: Optical Correction — Glasses prescribed at investigator discretion
  Arms: Continued Optical Correction Group

SUMMARY:
Participants eligible for the study will be randomly allocated (1:1:1) to receive either Luminopia dichoptic treatment while wearing optical correction if needed, Vivid Vision dichoptic treatment while wearing optical correction if needed, or continued optical correction alone if needed, with clinical assessments at 9- and 18-weeks post-randomization.

At the 18-week primary outcome visit, participants who were randomly assigned to receive optical correction alone if needed with an IOD of 1 logMAR line (5 letters) or more, will be offered randomization to Luminopia or Vivid Vision dichoptic therapy and if they accept, followed forward with visits at 27- and 36-weeks post-randomization.

The study will end for all other participants at 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 to <13 years.
2. VA, measured in each eye without cycloplegia in current refractive correction (if applicable) using the E-ETDRS VA protocol on a study-approved device displaying single surrounded optotypes, as follows:

   1. VA in the amblyopic eye 20/40 to 20/200 inclusive (33 to 72 letters with E-ETDRS).
   2. VA in the fellow eye 20/25 or better (≥ 78 letters with E-ETDRS).
   3. Interocular difference ≥ 3 logMAR lines (≥ 15 letters) i.e., amblyopic eye VA at least 3 logMAR lines worse than fellow eye VA).
3. Amblyopia associated with strabismus, anisometropia, or both (previously treated or untreated).

   1. Criteria for strabismic amblyopia: At least one of the following must be met:

      * Presence of a heterotropia on examination at distance or near fixation (with optical correction), must be <=5 prism diopters (∆) by SPCT at distance and near fixation.
      * Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia).
   2. Criteria for anisometropia: At least one of the following criteria must be met:

      * ≥1.00 D difference between eyes in spherical equivalent (SE).
      * ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes.
   3. Criteria for combined-mechanism: Both of the following criteria must be met:

      * A criterion for strabismus is met (see above).
      * ≥1.00 D difference between eyes in SE OR ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes.
4. No more than 2 weeks (cumulative) of prior dichoptic treatment
5. No treatment with cycloplegic eyedrops (e.g., atropine) in the past 2 weeks; other treatments allowed up to enrollment but then must be discontinued.
6. Refractive correction is required (single vision lenses or contact lenses) for any of the following refractive errors based on a cycloplegic refraction completed within the last 7 months:

   * Hypermetropia of 2.50 D or more by SE
   * Myopia of amblyopic eye of 0.50D or more SE
   * Astigmatism of 1.00D or more
   * Anisometropia of more than 0.50D SE

   NOTE: Children with cycloplegic refractive errors that do not fall within the requirements above for refractive correction may be given refractive correction at investigator discretion but must follow the study-specified prescribing guidelines, as detailed below.

   NOTE: Monocular or binocular contact lens wear is allowed provided the contact lenses meet the refractive error correction requirements below. For each child, all testing must be performed using the same form of optical correction (i.e., no changing between contacts and spectacles).
   1. Spectacles/contact lens correction prescribing instructions referenced to the cycloplegic refraction completed within the last 7 months:

      * SE must be within 0.50D of fully correcting the anisometropia (if new glasses are prescribed, reduction in plus sphere must be symmetric in the two eyes).
      * SE must not be under corrected by more than 1.50D SE.
      * Cylinder power in both eyes must be within 0.50D of fully correcting the astigmatism.
      * Axis must be within +/- 10 degrees if cylinder power is ≤1.00D, and within +/- 5 degrees if cylinder power is >1.00D.
      * Myopia must not be under corrected by more than 0.25D or over corrected by more than 0.50D SE, and any change must be symmetrical in the two eyes.
   2. Spectacles/contact lens correction (with or without other treatment such as patching) meeting the above criteria must be worn:

      * For at least 18 weeks OR until VA stability is documented (defined as <1-line change by the same testing method measured on 2 consecutive exams at least 9 weeks apart).
      * For determining VA stability (non-improvement):

        * The first of two measurements may be made 1) in current correction, or 2) in trial frames with or without cycloplegia or 3) without correction (if new correction is prescribed),
        * The second measurement must be made without cycloplegia in the correct spectacles/contact lens correction that has been worn for at least 9 weeks.
        * NOTE: Because this determination is a pre-randomization, the method of measuring VA is not mandated.
7. Participant is willing to wear a headset.
8. Participant is willing to continue full-time spectacles/contact lens wear (if needed).
9. Interpupillary distance of 52mm to 72mm inclusive.
10. Investigator is willing to prescribe continued spectacles/contact lens correction (if needed) or either dichoptic device per protocol.
11. Participant is willing to accept assignment to either continued spectacles/ contact lens wear alone, dichoptic movies/shows (view 1 hour per day 6 days per week) OR dichoptic games (play approximately 25 minutes per day, 6 days per week) for 19 weeks.
12. Parent understands the protocol and is willing to accept randomization.
13. Parent has phone (or access to phone) and is willing to be contacted by JAEB Center staff.
14. Relocation outside of area of an active PEDIG site for this study within the next 36 weeks is not anticipated.

Exclusion Criteria:

1. Heterotropia more than 5∆ at distance or near (measured by SPCT in current correction)
2. Prism greater than a total of 8 diopters horizontal and 1 diopter vertical in the refractive correction at time of enrollment.
3. Current bifocal spectacles (eligible only if bifocal discontinued 2 weeks prior to enrollment).
4. Myopia greater than -6.00D spherical equivalent in either eye.
5. Ocular co-morbidity that may reduce VA determined by an ocular examination performed within the past 7 months (Note: nystagmus per se does not exclude the participant if the above visual acuity criteria are met using patch occlusion. Fogging is not permitted).
6. Diplopia more than once per week over the last week prior to enrollment by parental report.
7. History of light-induced seizures.
8. Known simulator sickness.
9. Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Participants with mild speech delay or reading and/or learning disabilities are not excluded.
10. Immediate family member (biological or legal guardian, child, sibling, parent) of investigative site personnel directly affiliated with this study or an employee of the JAEB center for Health Research.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 252 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in amblyopic eye logMAR distance VA | 18 Weeks
  between randomization and 18 weeks

SECONDARY OUTCOMES:
Functional Vision, Social, and Frustration/Worry quality of life domains as measured by the Pediatric Eye Questionnaire (PedEyeQ). | 18 Weeks
  Questionnaire outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marjean T Kulp, OD, Study Chair — Ohio State University; Benajmin G Jastrzembski, MD, Study Chair — University of California, Davis
Locations (58):
- United States (58):
  - UAB Pediatric Eye Care; Birmingham Health Care, Birmingham, Alabama
  - Midwestern University Eye Institute, Glendale, Arizona
  - Phoenix Children's Medical Group - Ophthalmology, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Arkansas Childrens, Little Rock, Arkansas
  - McFarland Eye Care Center, Little Rock, Arkansas
  - University Eye Center at Ketchum Health, Anaheim, California
  - Univ. of California- Berkeley, Berkeley, California
  - Univ of California, Irvine- Gavin Herbert Eye Institute, Irvine, California
  - Stanford University, Palo Alto, California
  - Western University College of Optometry, Pomona, California
  - University of California, Davis, Sacramento, California
  - University of California San Francisco Department of Ophthalmology, San Francisco, California
  - Nova Southeastern University College of Optometry, The Eye Institute, Fort Lauderdale, Florida
  - University of South Florida (USF) Eye, Tampa, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - Midwestern University Eye Institute, Downers Grove, Illinois
  - Progressive Eye Care, Lisle, Illinois
  - Indiana School of Optometry, Bloomington, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Dept of Ophthalmology, Prairie Village, Kansas
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Wilmer Eye Institute, Baltimore, Maryland
  - New England College of Optometry, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston Children's Hospital Waltham, Boston, Massachusetts
  - Michigan College of Optometry at Ferris State Univ, Big Rapids, Michigan
  - Pediatric Ophthalmology, P.C., Grand Rapids, Michigan
  - Zenith Vision Development Center, Duluth, Minnesota
  - University of Minnesota-Minnesota Lions Children's Eye Clinic, Minneapolis, Minnesota
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - PineCone Vision Center, Sartell, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - State University of New York, College of Optometry, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - University of North Dakota, Grand Forks, North Dakota
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cole Eye Institute, Cleveland, Ohio
  - Ohio State University College of Optometry, Columbus, Ohio
  - Rainbow Babies and Children's Hospital Dept of Ophth, Mayfield Heights, Ohio
  - River View Family Eyecare, Albany, Oregon
  - OHSU Casey Eye Institute, Portland, Oregon
  - Pediatric Ophthalmology of Erie, Erie, Pennsylvania
  - Conestoga Eye, Lancaster, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Salus University/Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - Storm Eye Institute, Mt. Pleasant, South Carolina
  - Southern College of Optometry, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Houston - College of Optometry, Houston, Texas
  - University of Houston College of Optometry, Houston, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Virginia Pediatric Eye Center, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the Pediatric Eye Disease Investigator Group (PEDIG) public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after publication.
Access Criteria: Users accessing the data must enter an email address
URL: http://pedig.jaeb.org

DOCUMENTS (3):
  • Study Protocol (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT06524882/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT06524882/SAP_001.pdf
  • Informed Consent Form (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT06524882/ICF_002.pdf